CLINICAL TRIAL: NCT00452348
Title: A 52-week, Randomized, Double-Blind, Parallel-Group Study of Fluticasone Propionate/Salmeterol DISKUS Combination Product (FSC) 250/50 mcg BID and Fluticasone Propionate (FP) DISKUS 250 mcg BID in Treatment of Subjects With Asthma
Brief Title: A 12-Month Study Comparing Fluticasone Propionate/Salmeterol (ADVAIR) DISKUS Combination Product 250/50mcg Twice Daily To Fluticasone Propionate (FLOVENT) DISKUS 250 mcg Twice Daily In Symptomatic Patients With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADA109057
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: FLOVENT; fluticasone; 12 month; salmeterol; asthma; ADVAIR
MeSH Terms: conditions — Asthma | interventions — Fluticasone; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fluticasone propionate 250 mcg BID (Active Comparator): Fluticasone propionate 250 mcg BID
  Interventions: Drug: Fluticasone propionate 250 mcg BID
- Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID (Active Comparator): Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID
  Interventions: Drug: Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID

INTERVENTIONS:
Drug: Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID — Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID
  Other Names: Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID and Fluticasone propionate 250 mcg BID
  Arms: Fluticasone Propionate/salmeterol xinofoate 250/50 mcg BID
Drug: Fluticasone propionate 250 mcg BID — Fluticasone propionate 250 mcg BID
  Arms: Fluticasone propionate 250 mcg BID

SUMMARY:
This purpose of this study is to show the superiority and long term safety and efficacy of adding a long acting beta agonist (salmeterol) to constant dose of an inhaled corticosteroid (fluticasone propionate) in symptomatic subjects with asthma. The 12-month assessment of asthma control will provide key information on the efficacy and safety of the combination therapy. The safety measure will be an assessment of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for enrollment in the study must meet all of the following criteria:

  1. Consent: A signed and dated written informed consent must be obtained from the subject and/or subject's legally acceptable representative prior to study participation.
  2. Type of Subject: Outpatient
  3. Gender: Male or female Females are eligible to participate only if they are currently non-pregnant and non-lactating.

A female is eligible to enter and participate in the study if she is:

1. of non-child-bearing potential; OR
2. of child-bearing potential but has a negative urinary pregnancy test at Screening (Visit 1 and when specified in Appendix 1) and agrees to take contraceptive precautions (including abstinence) which are adequate to prevent pregnancy during the study.

   Acceptable methods of contraception [Hatcher, 2004] are:

   - Abstinence
   * oral contraceptive (either combined or progestogen only)
   * injectable progestogen
   * implants of levonorgestrel
   * estrogenic vaginal ring
   * percutaneous contraceptive devices
   * intrauterine device (IUD) or intrauterine system (IUS) with published data showing that the lowest expected failure rate is less than 1% per year
   * male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study and is the sole sexual partner for that female subject
   * double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent

     1. Age: A subject must be 12 years of age at Visit 1 (screening).
     2. Asthma Diagnosis: A documented diagnosis of persistent asthma, for at least six months, as defined by the following American Thoracic Society definition:

   Asthma is a clinical syndrome characterized by increased responsiveness of the airways to a variety of stimuli. The major symptoms of asthma are episodes of dyspnea, wheezing, and cough, which may vary from mild and almost undetectable to severe and unremitting (status asthmaticus). The primary physiological manifestation of this hyperresponsiveness is variable airway obstruction. This can take the form of spontaneous fluctuations in the severity of obstruction, substantial improvements in the severity of obstruction following bronchodilators or corticosteroids, or increased obstruction caused by drugs or other stimuli [American Thoracic Society, 1987].
   1. Asthma Medication History: A subject must be using a low to medium dose of an ICS (Table 1) OR a combination of controller medications (Table 2), containing a low (total daily) dose ICS (as defined in Table 1) for at least 4 weeks preceding screening.

   Table 1 (ICS Dosage Table) Inhaled Corticosteroid (Dosage (mcg/day))(LowMedium) Beclomethasone dipropionate CFC (168 = 504> 504 = 840) Beclomethasone dipropionate HFA (80 = 240>240 = 640) Triamcinolone acetonide (400 = 1000>1000 = 2000) Flunisolide (500 = 1000> 1000 = 2000) Fluticasone propionate inhalation aerosol (176 = 220> 220 = 440) Fluticasone propionate inhalation powder (100 = 250> 250 = 500) Budesonide1 (200 = 600> 600 =1200) Mometasone (200 = 400> 400 = 800) Ciclesonide (80 = 160>160 = 320)

   1.Respules are allowed at a dosage of 250-500mcg/day.

   Table 2 (Asthma Controller Medications) Asthma Controller Medication(s) Low dose ICS + Leukotriene modifiers Low dose ICS + Theophylline products Low Dose ICS + Inhaled anticholinergics or combination products (e.g., Atrovent or Combivent) Low Dose ICS + Long acting inhaled anticholinergic (e.g. Spiriva) Low dose ICS+ long acting beta agonist or combination products containing a low dose ICS and a long-acting beta-agonists (e.g. ADVAIR™/SERETIDE™1 100/50 mcg BID or Symbicort 160/9 mcg BID (i.e 80/4.5 mcg two inhalations BID)

   1.ADVAIR/SERETIDE =250/50 mcg BID or Symbicort 320/9 mcg BID (i.e 160/4.5 mcg two inhalation BID) are not permitted.
   1. Pulmonary function: A pre-albuterol (salbutamol) FEV1 of 50% and 85% of predicted normal value at screening (Visit 1) after withholding asthma medications as detailed in the protocol (Section 6.8.1). Predicted FEV1 will be based on the National Health and Nutrition Examination Survey (NHANES III) predicted normal values for ages 8 years and older [Hankinson, 1999].
   2. Reversibility: An increase in FEV1 of 12% over the pre-albuterol (salbutamol) FEV1 within 30 minutes after the inhalation of 2-4 puffs of albuterol (salbutamol). Historical documentation of reversibility will not be permitted.
   3. Asthma symptom criteria: Each subject must have experienced asthma symptoms requiring albuterol (salbutamol) use within the 4 weeks preceding screening (Visit 1).

   Specific information regarding warnings, precautions, contraindications, adverse events, and other pertinent information on the investigational product that may impact subject eligibility is provided in the IB and the product labels.

   Exclusion Criteria:
   * Subjects meeting any of the following criteria must not be enrolled in the study:

     1.Life-Threatening Asthma: A subject must not have life-threatening asthma. Life-threatening asthma is defined for this protocol as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, or hypoxic seizures, or asthma-related syncopal episode(s) within the 12 months prior to screening (Visit 1).

     2.Worsening of Asthma: A subject must not have experienced a worsening of asthma which involved an ER visit, hospitalization or use of oral/parenteral corticosteroids within 4 weeks of screening (Visit 1).

     3.Intermittent, Seasonal, or Exercise-Induced Asthma Alone: Subjects with only intermittent or seasonal or exercise-induced asthma are excluded from participation in this study.

     4.Concurrent Respiratory Disease: A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.

     5.Concurrent Conditions/Diseases: A subject with historical or current evidence of any clinically significant, co-morbid or uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbated during the study.

   The list of excluded conditions/diseases includes, but is not limited to:

   congestive heart failure known aortic aneurysm clinically significant coronary clinically significant cardiac arrhythmia heart disease stroke within 3 months of screening (Visit 1) uncontrolled hypertension coronary artery disease hematologic, hepatic, or renal disease cystic fibrosis poorly controlled peptic ulcer dyspnea by any other cause than asthma gastroesophageal reflux disease (GERD) not controlled by pharmacotherapy and may be causing/contributing to subject's respiratory symptoms thyrotoxicosis hypokalemia immunologic compromise current malignancy1 tuberculosis (current or quiescent) Cushing's or Addison's disease pneumonia, pneumothorax, chronic bronchitis or atelectasis uncontrolled diabetes mellitus recent history of drug or alcohol abuse 1.history of malignancy is acceptable only if subject has been in remission for one year prior to screening (Visit 1; remission = no treatment for the malignancy in the 12 months prior to screening [Visit 1])
   1. Drug Allergy: A subject must not have had any immediate or delayed hypersensitivity to any beta2-agonist; sympathomimetic drug; any intranasal; inhaled or systemic corticosteroid therapy; lactose; or have a severe milk protein allergy.
   2. Respiratory Tract Infections: A subject must not have had any sinus, middle ear, oropharyngeal, upper or lower respiratory tract infection symptoms that have not resolved at least 7 days immediately preceding screening (Visit 1).
   3. Asthma Medications: Asthma medications listed below must not have been used prior to screening (Visit 1) for the required exclusion period as indicated below:

      Medication (Exclusion Period Prior to screening (Visit 1)) Oral or parenteral systemic corticosteroids (4 weeks) Omalizumab (Xolair) (6 months)

   <!-- -->

   1. Concurrent Medications: A subject must not have the concurrent use of any of the following medications that interact with any of the study drugs used in this study, or that may affect the course of asthma or interact with sympathomimetic amines, such as:

      - beta-adrenergic receptor blocking agents

      - monoamine oxidase (MAO) inhibitors

      - tricyclic antidepressants

      - ritonavir
      * ketoconazole
   2. Concurrent use of asthma medications: Concurrent use of all asthma medications (other than protocol defined study and rescue medications and oral/parenteral corticosteroids) are prohibited during the study.
   3. Concomitant use of leukotriene modifiers (LTM) for allergies is prohibited. A subject must not be on LTM for treatment of nasal allergies that requires regular maintenance therapy. Substitution with any other antihistamine is permitted.
   4. Immunosuppressive Medications: A subject must not be using, or require the use of, immunosuppressive medications during the study.
   5. Immunotherapy for the treatment of allergies is not allowed during the study unless the subject has used a constant dose for 4 weeks prior to Screening (Visit 1) and the same dose will be continued throughout the study.
   6. Tobacco Use: >10 pack year history or use of any tobacco products within 1 year of screening (Visit 1). This includes cigarettes, cigars, pipe, chewing tobacco, and snuff.
   7. Questionable Validity of Consent: A subject must not have any infirmity or disability that would limit the subject's consent.
   8. Positive Pregnancy Test (for all females who have had menarche): A current positive pregnancy test.
   9. Investigational Medications: A subject must not have had use of any investigational drug within 30 days of screening (Visit 1).
   10. Site Affiliation: A subject may not participate if he/she is a participating investigator, sub-investigator, study coordinator, employee of a participating investigator or is in any way associated with the administration of the study. Immediate family members of these individuals are also excluded.
   11. Compliance with Study Requirements: A subject may not participate if, in the opinion of the investigator, there are present or anticipated circumstances that will prohibit the subject from being compliant with study visits and procedures (e.g. geographic location that will prohibit subject from required clinic visit schedule).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (78):
- United States (57):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Pueblo, Colorado
  - GSK Investigational Site, Hudson, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Collegeville, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (6):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
- Brazil (5):
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Florianópolis, Santa Catarina
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (9):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Saint-Léonard, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- GSK Investigational Site, Quezon City, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Anderson WH, Koshy BT, Huang L, Mosteller M, Stinnett SW, Condreay LD, Ortega H. Genetic analysis of asthma exacerbations. Ann Allergy Asthma Immunol. 2013 Jun;110(6):416-422.e2. doi: 10.1016/j.anai.2013.04.002. PMID 23706709
- [Background] Kerwin E, Prazma CM, Sutton L, Stempel DA. Safety and efficacy of long-term treatment with fluticasone propionate and salmeterol via DISKUS versus fluticasone propionate alone. Clin Res Reg Aff 2011;28(1):14-21.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ADA109057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- FSC DISKUS 250/50 mcg BID: Fluticasone Propionate/Salmeterol DISKUS Combination Product (FSC) 250/50 micrograms (mcg) twice daily (BID) for 52 weeks
- FP DISKUS 250 mcg BID for 52 Weeks: Fluticasone Propionate (FP) DISKUS 250 mcg BID for 52 weeks
Period: Overall Study
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks
Started | 310 | 318
Completed | 231 | 234
Not Completed | 79 | 84
Not completed — Adverse Event | 6 | 9
Not completed — Lack of Efficacy | 10 | 9
Not completed — Lost to Follow-up | 14 | 8
Not completed — Protocol Violation | 22 | 28
Not completed — Withdrawal by Subject | 18 | 21
Not completed — Other | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks | Total
Number analyzed (Participants) | 310 | 318 | 628
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.71) | 39.6 (16.56) | 40.2 (16.15)
Gender [Count of Participants; unit: Participants]
  Female | 186 | 181 | 367
  Male | 124 | 137 | 261
Race/Ethnicity, Customized [Number; unit: participants]
  White | 254 | 262 | 516
  African American | 29 | 27 | 56
  Asian | 20 | 25 | 45
  American Indian | 2 | 0 | 2
  Other | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Pre-dose FEV1 Over Weeks 1-52
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), which is the volume of air exhaled from the lungs in one second. Change from baseline was calculated as the average of the Week 1 through Week 52 values minus the baseline value.
Time Frame: Baseline and Week 1 through Week 52
Population: Intent-to-Treat (ITT) Population: all participants randomized to study drug who had at least one on-treatment FEV1
Measure: Mean (Standard Error); unit: Liters
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks
Number analyzed (Participants) | 303 | 304
Liters | 0.16 (0.017) | 0.12 (0.020)
Statistical Analysis 1: Comparison: FSC DISKUS 250/50 mcg BID vs FP DISKUS 250 mcg BID for 52 Weeks; Test type: Superiority or Other; p = 0.090, ANCOVA; Least Squares Mean = 0.04, 95% CI [-0.01 to 0.09]

2. Secondary Outcome: Mean Change From Baseline in AM PEF Over Weeks 1-52
Description: Morning (AM) peak expiratory flow (PEF) is defined as the maximum volume of air exhaled in liters per minute. Change from baseline was calculated as the average of the Week 1 through Week 52 values minus the baseline value.
Time Frame: Baseline and Week 1 through Week 52
Population: Participants in the ITT Population who had a minimum of 1 week PEF values
Measure: Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks
Number analyzed (Participants) | 305 | 310
Liters/minute (L/min) | 27.7 (2.85) | 14.6 (2.49)

3. Secondary Outcome: Mean Change From Baseline in the Percentage of Symptom-free Days Over Weeks 1-52
Description: A symptom-free day was defined as a day without asthma symptoms, as measured via the daily asthma symptom score (measuring symptoms during the day and previous night) on a 6-point scale (ranging from 0 to 5). A symptom score of 0=no symptoms, 1=symptoms for one short period, 2=symptoms for two or more short periods, 3=symptoms that did not affect normal daily activities, 4=symptoms that did affect normal daily activities, 5=symptoms so severe that daily activities could not be performed. Change from baseline was calculated as the average of the Week 1-Week 52 values minus the baseline value.
Time Frame: Baseline and Week 1 through Week 52
Population: Participants in the ITT Population for which at least 1 week of diary data were provided
Measure: Mean (Standard Error); unit: Percentage of symptom-free days
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks
Number analyzed (Participants) | 305 | 310
Percentage of symptom-free days | 37.4 (2.03) | 28.9 (1.82)

4. Secondary Outcome: Rate of Asthma Attacks Per Participant Per Year
Description: The rate of asthma attacks was defined as the mean number of attacks per participant per year. An asthma attack was defined as a >=20% decrease in AM PEF, a >=70% increase in albuterol use, or the occurrence of an asthma exacerbation requiring oral steroids or hospitalization.
Time Frame: Week 1 through Week 52
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: attacks per participant per year
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks
Number analyzed (Participants) | 310 | 318
attacks per participant per year | 2.63 [2.17 to 3.19] | 2.73 [2.26 to 3.31]

ADVERSE EVENTS:
Arm/Group | FSC DISKUS 250/50 mcg BID | FP DISKUS 250 mcg BID for 52 Weeks
Serious Adverse Events (participants affected / at risk) | 7/310 | 9/318
Other Adverse Events (participants affected / at risk) | 184/310 | 201/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DISKUS 250/50 mcg BID (N=310) | FP DISKUS 250 mcg BID for 52 Weeks (N=318)
Cardiac death (General disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Breast cancer (Reproductive system and breast disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC DISKUS 250/50 mcg BID (N=310) | FP DISKUS 250 mcg BID for 52 Weeks (N=318)
Upper respiratory tract infection (Infections and infestations) | 45 | 55
Nasopharyngitis (Infections and infestations) | 54 | 70
Bronchitis (Infections and infestations) | 34 | 38
Influenza (Infections and infestations) | 15 | 21
Sinusitis (Infections and infestations) | 33 | 40
Headache (Nervous system disorders) | 51 | 60
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 19
Rhinitis (Infections and infestations) | 23 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.